CLINICAL TRIAL: NCT05267171
Title: Effect of an Educational Intervention for the Prevention of Breast Cancer by Modifying Risk Behaviors Through the Use of a Web-app: Project Breast47
Brief Title: Project Breast47: Effect of an Educational Intervention
Acronym: Breast47
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Claudia Leirós, RN; MSC, University of Oviedo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021.341
Record Dates: First submitted 2022-02-03; First posted 2022-03-04 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Breast Neoplasm; Primary Prevention; Risk Factors; Telemedicine
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Web access
- Control group (No Intervention)

INTERVENTIONS:
Other: Web access — The intervention group will have access to the website where the information is provided. The control group will not have this access.
  Arms: Intervention group

SUMMARY:
Breast cancer is the most frequently diagnosed malignant tumor in women. In 2018, in Spain, the estimated incidence was 101/100,000 women.

Screening strategies and greater knowledge of risk factors by the population have contributed to a better prognosis. Specifically, in the case of behavioral factors, making women aware of their influence enables them to establish preventive measures themselves.

Technologies are becoming a channel of communication, from a healthcare perspective, between the population and healthcare personnel. There are even specific terms like eHealth or mHealth. There is beginning to be evidence that collects the benefits and ways of using web-apps to achieve modification of risky behaviors and/or behaviors to prevent pathologies are acquired.

The use of digital media, such as a web-app, to publicize BC risk factors makes it possible to specifically establish measures aimed at reducing its prevalence, which in turn will contribute to reducing the number of cases of BC. CM.

On the other hand, making women aware of their BC risk factors, as well as quantifying the risk of developing the tumor, is useful for them to become aware of the magnitude of the problem and adopt measures to minimize their risk.

Since there is no digital strategy in Asturias that informs and reduces the risk of developing breast cancer, through the modification of the main risk factors, in young women, the present study has been proposed with the aim of evaluating the effectiveness and feasibility of an educational intervention for BC risk prevention through the use of a Web-App in women residing in health area VII of the Principality of Asturias.

ELIGIBILITY:
Inclusion Criteria:

* Women who agree to participate with no previous diagnosis of breast cancer

Exclusion Criteria:

* Women who do not have adequate physical or psychological characteristics to participate in the study
* Women who do not have the means to regularly access the web-app that will be used to develop the educational intervention
* Women who cannot be contacted by email

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 451 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Leirós, Principal Investigator — Universidad de Oviedo
Locations (1):
- Universidad de Oviedo, Oviedo, Principality of Asturias, Spain

REFERENCES:
- [Derived] Martin-Payo R, Leiros-Diaz C, Urena-Lorenzo A, Cachero-Rodriguez J, Fernandez-Arce L, Fernandez-Alvarez MDM. A web-based intervention to promote healthy lifestyles in women under 45 years: a randomized controlled trial (RCT) for breast cancer prevention. Mhealth. 2025 Oct 28;11:54. doi: 10.21037/mhealth-25-2. eCollection 2025. PMID 41211018

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: The control group will not have this access.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 207 | 244
Completed | 101 | 188
Not Completed | 106 | 56

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Web access: The intervention group will have access to the website where the information is provided.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 207 | 244 | 451
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.88 (5.56) | 38.76 (5.28) | 38.82 (5.36)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Women | 207 | 244 | 451
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Civil Status [Count of Participants; unit: Participants]
  Single | 50 | 60 | 110
  Separated, divorced or widowed | 10 | 4 | 14
  Married or in a relationship | 147 | 180 | 327
Educational level [Count of Participants; unit: Participants]
  Primary studies | 6 | 2 | 8
  Secondary studies | 17 | 16 | 33
  High school studies | 21 | 24 | 45
  University studies | 101 | 129 | 230
  Others | 62 | 73 | 135
Employment [Count of Participants; unit: Participants]
  Employed | 171 | 213 | 384
  Unemployed | 36 | 31 | 67
Family history of cancer [Count of Participants; unit: Participants]
  Yes | 152 | 177 | 329
  No | 55 | 67 | 122
History of breast cancer in the family [Count of Participants; unit: Participants]
  Yes | 67 | 86 | 153
  No | 140 | 158 | 298

OUTCOME MEASURES:

1. Primary Outcome: Behavioral BC Risk With an Educational Intervention for Prevention
Description: The information related to the behavioral will be evaluated with the Motiva.Diaf questionnaire.
  The questionnaire allows you to evaluate adherence to healthy recommendations. This includes 12 multiple choice questions related to diet (questions 1 to 7) and physical activity (questions 8 to 12). Each is expressed dichotomously (follow this recommendation/do not follow this recommendation).
  Finally, the quantitative variable adherence to healthy recommendations is created as a result of the score of each of the items in its dichotomous interpretation, with a range from 0 (worst adherence to healthy recommendations) to 12 (greatest adherence to healthy recommendations).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 207 | 244
units on a scale | 8.10 (2.57) | 8.15 (2.60)

2. Primary Outcome: Feasibility of an Educational Intervention for BC Risk Prevention Through the Use of a Web-App
Description: PostIntervention - Feasibility will be measured with satisfaction questionnaire.
  Satisfaction related to the web-app used in the intervention was measured with the SUS scale in its validated version in Spanish. This is a standardized scale that allows measuring the perception of the usability and satisfaction of a system.
  It consists of 10 items that are scored on a Likert-type scale ranging from 1, which is totally disagree, to 5, which is totally agree.
  After calculating the result, we will obtain a score in a range from 0 to 100, where its average is 68. Above this figure and up to 84, it is considered "good usability." Equal to or greater than 85 is considered "excellent usability".
  This part was only evaluated in those women belonging to the intervention group and who, therefore, had been able to use the web-app.
Time Frame: 12 weeks (end of intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 101
units on a scale | 71.87 (17.94)

3. Primary Outcome: Knowledge of BC Risk With an Educational Intervention for Prevention
Description: Knowledge of risk factors and signs of BC with the MARA questionnaire. This questionnaire consists of 4 subscales and a total of 31 items, of which 9 are related to knowledge of risk factors and 9 to signs and symptoms.
  The items related to knowledge about risk factors are aimed at both modifiable factors (4 items) and non-modifiable factors (5 items). Each success adds 1 and each failure adds 0, so the range of modifiable factors is 0 to 4 and non-modifiable factors is 0 to 5. The items on knowledge of signs and symptoms address both the specific ones (4 items) as non-specific ones (5 items). In the same way as the previous one, in this section the successes add up to 1 and the failures add up to 0. The range, therefore, of the specific ones is from 0 to 4 and of the non-specific ones is from 0 to 5. The total score range for both Risk as for signs and symptoms is between 0 and 9, with 0 being the maximum error or lack of knowledge and 9 being the maximum success or knowledge.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 207 | 244
units on a scale | 4.61 (2.01) | 4.65 (2.04)

4. Primary Outcome: Barriers to Prevent BC With an Educational Intervention for Prevention
Description: Barriers to prevent BC with the MARA questionnaire. This questionnaire consists of 4 subscales and a total of 31 items, of which 7 items are perceived barriers to carrying out prevention strategies.
  The score is represented on a Likert-type scale with a range from 1 (totally disagree) to 5 (totally agree), with the total score of perceived barriers being between 7 and 35 points (the lower the score, the fewer the perceived barriers).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 207 | 244
units on a scale | 28.60 (3.70) | 28.77 (4.03)

5. Primary Outcome: BC Risk Perception With an Educational Intervention for Prevention
Description: Risk perception with the MARA questionnaire. This questionnaire consists of 4 subscales and a total of 31 items, of which 6 items relate to the perception of risk of developing breast cancer.
  The score is represented on a Likert-type scale with a range from 1 (totally disagree) to 5 (totally agree), with the total risk perception score being between 6 and 30 points (the lower the score, the lower the risk perception).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 207 | 244
units on a scale | 11.34 (2.89) | 11.22 (3.04)

6. Primary Outcome: Breast Self-examination With an Educational Intervention for Prevention
Description: Carrying out self-examination through objective questioning. To find out whether self-examination was performed, a question was asked: "Do you perform breast self-examination once a month?" with a dichotomous yes/no response option.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 207 | 244
Participants
  Breast self-examination | 123 | 142
  No breast self-examination | 84 | 102

7. Primary Outcome: Knowledge of BC Risk With an Educational Intervention for Prevention
Description: Post Intervention - Risk perception with the MARA questionnaire. This questionnaire consists of 4 subscales and a total of 31 items, of which 6 items relate to the perception of risk of developing breast cancer.
  The score is represented on a Likert-type scale with a range from 1 (totally disagree) to 5 (totally agree), with the total risk perception score being between 6 and 30 points (the lower the score, the lower the risk perception).
Time Frame: 12 weeks (end of intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 101 | 188
units on a scale | 10.19 (3.07) | 11.11 (3.14)

8. Primary Outcome: Behavioral BC Risk With an Educational Intervention for Prevention
Description: PostIntervention - The information related to the behavioral will be evaluated with the Motiva.Diaf questionnaire.
  The questionnaire allows you to evaluate adherence to healthy recommendations. This includes 12 multiple choice questions related to diet (questions 1 to 7) and physical activity (questions 8 to 12). Each is expressed dichotomously (follow this recommendation/do not follow this recommendation).
  Finally, the quantitative variable adherence to healthy recommendations is created as a result of the score of each of the items in its dichotomous interpretation, with a range from 0 (worst adherence to healthy recommendations) to 12 (greatest adherence to healthy recommendations).
Time Frame: 12 weeks (end of intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 101 | 188
units on a scale | 9.21 (2.20) | 8.40 (2.59)

9. Primary Outcome: Knowledge for BC Risk With an Educational Intervention for Prevention
Description: PostIntervention - Knowledge of risk factors and signs of BC with the MARA questionnaire (4 subscales and 31 items of which 9 are related to knowledge of risk factors and 9 to signs and symptoms) The items related to knowledge about risk factors are aimed at both modifiable factors (4 items) and non-modifiable factors (5 items). Each success adds 1 and each failure adds 0, so the range of modifiable factors is 0 to 4 and non-modifiable factors is 0 to 5. The items on knowledge of signs and symptoms address both the specific ones (4 items) as non-specific ones (5 items). In the same way as the previous one, in this section the successes add up to 1 and the failures add up to 0. The range, therefore, of the specific ones is from 0 to 4 and of the non-specific ones is from 0 to 5. The total score range for both Risk as for signs and symptoms is between 0 and 9, with 0 being the maximum error or lack of knowledge and 9 being the maximum success or knowledge.
Time Frame: 12 weeks (end of intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 101 | 188
units on a scale | 5.87 (1.71) | 5.13 (1.97)

10. Primary Outcome: Barriers to Prevent BC With an Educational Intervention for Prevention
Description: PostIntervention - Barriers to prevent BC with the MARA questionnaire. This questionnaire consists of 4 subscales and a total of 31 items, of which 7 items are perceived barriers to carrying out prevention strategies.
  The score is represented on a Likert-type scale with a range from 1 (totally disagree) to 5 (totally agree), with the total score of perceived barriers being between 7 and 35 points (the lower the score, the fewer the perceived barriers).
Time Frame: 12 weeks (end of intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 101 | 188
units on a scale | 29.59 (3.68) | 28.88 (4.24)

11. Primary Outcome: Breast Self-examination With an Educational Intervention for Prevention
Description: PostIntervention - Carrying out self-examination through objective questioning. To find out whether self-examination was performed, a question was asked: "Do you perform breast self-examination once a month?" with a dichotomous yes/no response option.
Time Frame: 12 weeks (end of intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 101 | 188
Participants
  Breast self-examination | 83 | 122
  No breast self-examination | 18 | 66

ADVERSE EVENTS:
Time Frame: In this project, adverse event were not collected.
Description: In this project, adverse event were not collected, what explains why the number of participants at risk for Serious Adverse Events and risk for All-Cause Mortality is zero
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT05267171/Prot_SAP_ICF_000.pdf